CLINICAL TRIAL: NCT04914013
Title: Invasive Fungal Sinusitis Among Post COVID-19 Survivors in Upper Egypt
Brief Title: Fugal Infection in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maiada K. Hashem, Lecturer, Assiut University
Other Study IDs: Fungi in COVID-19
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19, invasive fungal infection
MeSH Terms: conditions — COVID-19; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Screening early detection of invasive fungal sinusitis in COVID-19 positive patients

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2); the causative organism of Coronavirus disease 2019 (Covid-19); infects primarily the lungs leading to more than 100 million COVID-19 cases around the world, resulting in almost three million deaths. Covid-19 spectrum of symptoms expanded from upper respiratory tract infection to extensive viral pneumonia and respiratory failure. Covid-19 patients are highly susceptible to superimposed secondary infection especially fungal infections.

Acute invasive fungal sinusitis (AIFS) is one of the most aggressive forms of sinusitis that is commonly present in immunocompromised patients and frequently leads to significant mortality and morbidity. Mucormycosis a life threatening AIFS characterized by hyphal invasion and massive destruction of maxillofacial structures. Histological characters include mycotic infiltration of vessels with propensity to tissue infarction. In addition to other fungi such as Acinetobacter, Klebsiella, Enterobacter, Aspergillus and Candida that frequently lead to secondary fungal infection in Covid-19 patients.

The co-existence of Covid-19 and AIFS is due to immune dysregulation in Covid-19 patients as both CD4+ and CD8+ T lymphocytes are suppressed thus impair patients' innate immunity. In addition to the extensive use of steroids, broad spectrum antibiotics and monoclonal antibodies may contribute in fungal infection. Covid-19 patients with pre-existing conditions such as untreated HIV, organ transplantation, un controlled diabetes and malignancies are more susceptible to AIFS on the contrary Covid-19 patients with underlying chronic disease such as hypertension, chronic kidney and chronic heart disease usually are not associated with more risk of AIFS.

Taking in consideration raised incidence of morbidity and mortality associated with AIFS and on the other hand limited studies available especially in middle east region raised the importance of studying the incidence and the behaviour of AIFS in Covid-19 patients. This study aims to To assess the occurrence of AIFS superinfections in patients with Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with invasive fungal sinusitis, and are survivors of Covid19 infection, all cases diagnosed on the basis of the interim guidance of the World Health Organization (WHO) for diagnosis of SARS-CoV-2.

Exclusion Criteria:

* - Patients who received antifungal therapy within three days prior to sample collection.
* Patients refused to participate in the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with invasive fungal sinusitis, and are survivors of Covid19 infection, all cases diagnosed on the basis of the interim guidance of the World Health Organization (WHO) for diagnosis of SARS-CoV-2. Patients were recruited from:1- Otorhinolaryngology Department, Assuit university hospital. 2- Intermediate care unit of Internal Medicine department. 3-Respiratory Intensive care unite and chest department.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
detection of invasive fungal sinusitis after covid 19 infection. | baseline
  diagnosis of invasive fungal post COVID-19 infection

SECONDARY OUTCOMES:
Identify specific fungi that participate in IFS | 1 month
  specify by culture and sensitivity fungi that participate in invasive fungal sinusitis after covid 19 infection

REFERENCES:
- [Background] Fekkar A, Lampros A, Mayaux J, Poignon C, Demeret S, Constantin JM, Marcelin AG, Monsel A, Luyt CE, Blaize M. Occurrence of Invasive Pulmonary Fungal Infections in Patients with Severe COVID-19 Admitted to the ICU. Am J Respir Crit Care Med. 2021 Feb 1;203(3):307-317. doi: 10.1164/rccm.202009-3400OC. PMID 33480831
- [Background] Sharma S, Grover M, Bhargava S, Samdani S, Kataria T. Post coronavirus disease mucormycosis: a deadly addition to the pandemic spectrum. J Laryngol Otol. 2021 May;135(5):442-447. doi: 10.1017/S0022215121000992. Epub 2021 Apr 8. PMID 33827722
- [Background] Alanio A, Delliere S, Fodil S, Bretagne S, Megarbane B. Prevalence of putative invasive pulmonary aspergillosis in critically ill patients with COVID-19. Lancet Respir Med. 2020 Jun;8(6):e48-e49. doi: 10.1016/S2213-2600(20)30237-X. Epub 2020 May 20. No abstract available. PMID 32445626